CLINICAL TRIAL: NCT01738581
Title: Effectiveness of rTMS and Retraining in the Treatment of Focal Hand Dystonia
Brief Title: rTMS and Retraining in Focal Hand Dystonia
Acronym: DSS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0608M91226-2
Record Dates: First submitted 2012-09-18; First posted 2012-11-30 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Focal Dystonia
Keywords: focal hand dystonia (FHD); repetitive transcranial magnetic stimulation (rTMS); sensorimotor retraining
MeSH Terms: conditions — Dystonic Disorders; Dystonia, Focal, Task-Specific | interventions — Transcranial Magnetic Stimulation; Transcutaneous Electric Nerve Stimulation; Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rTMS + SMR, then rTMS + CTL (Experimental): First phase of treatment: Repetitive transcranial magnetic stimulation (rTMS) and sensorimotor retraining (SMR). Second phase of treatment: rTMS and control treatment (CTL) (CTL therapy consisted of non-specific therapy that includes stretching, massage, range of motion).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Behavioral: Sensorimotor Retraining; Behavioral: Non-specific Therapy
- rTMS + CTL, then rTMS + SMR (Experimental): First phase of treatment: Repetitive transcranial magnetic stimulation (rTMS) with non-specific therapy that includes stretching, massage, range of motion. Second phase of treatment: rTMS and sensorimotor retraining (SMR).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation; Behavioral: Sensorimotor Retraining; Behavioral: Non-specific Therapy

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Applied to the premotor cortex at 1 Hz at 90% resting motor threshold for 1200 pulses.
  Other Names: Magstim stimulator (Magstim Co. LTD, Whitland,UK); Neuromodulation
Behavioral: Sensorimotor Retraining — For sensorimotor retraining, a subset of the Learning-based Sensorimotor Training program was followed
  Other Names: Learning-based Sensorimotor Training program,; Sensory and motor Retraining
Behavioral: Non-specific Therapy — A non-specific massage and stretching program directed to the hand, wrist and forearm
  Other Names: Massage; Stretching

SUMMARY:
This study is exploring a new experimental procedure in dystonia called repetitive transcranial magnetic brain stimulation (TMS) combined with rehabilitation. The purpose of the study is to determine whether repetitive TMS is effective as a treatment to reduce symptoms in dystonia as demonstrated by improved motor performance.

DETAILED DESCRIPTION:
BACKGROUND: Though the etiology of focal hand dystonia (FHD) is uncertain, two primary factors implicated in the development of dystonic symptoms are excessive cortical excitability and impaired sensorimotor processing.

OBJECTIVE: The purpose of this study was to determine the functional efficacy and neural effects of a Dual intervention of rTMS and sensorimotor retraining. Our working hypothesis is: subjects receiving the combined intervention will (1) display significantly improved handwriting measures; (2) report significant improvement in daily functional ability; (3) display reduced hand cramping compared; and (4) demonstrate reduced corticospinal excitability after the Dual intervention when compared to the rTMS+ stretching and massage (Sham) intervention.

METHODS: A randomized, single-subject, multiple baseline design with crossover is used for this study that will examine ten subjects with FHD with two interventions: five days of low-frequency 1 Hz rTMS + sensorimotor retraining (Dual intervention) vs. rTMS + stretching and massage (Sham). The rTMS is applied to the premotor cortex at 1 Hz at 90% resting motor threshold for 1200 pulses. For sensorimotor retraining, a subset of the Learning-based Sensorimotor Training program was followed.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age
* Symptoms of focal hand dystonia or writer's cramp

Exclusion Criteria:

* History of seizure or other neurologic disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa J Kimberley, PhD, PT, Principal Investigator — University of Minnesota, Program in Physical Therapy
Locations (2):
- United States (2):
  - University of Minnesota, Program in Physical Therapy, Minneapolis, Minnesota
  - Program in Physical Therapy, University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Byl NN, Nagajaran S, McKenzie AL. Effect of sensory discrimination training on structure and function in patients with focal hand dystonia: a case series. Arch Phys Med Rehabil. 2003 Oct;84(10):1505-14. doi: 10.1016/s0003-9993(03)00276-4. PMID 14586919
- [Background] Kimberley TJ, Borich MR, Arora S, Siebner HR. Multiple sessions of low-frequency repetitive transcranial magnetic stimulation in focal hand dystonia: clinical and physiological effects. Restor Neurol Neurosci. 2013;31(5):533-42. doi: 10.3233/RNN-120259. PMID 23340117
- [Result] Kimberley TJ, Schmidt RL, Chen M, Dykstra DD, Buetefisch CM. Mixed effectiveness of rTMS and retraining in the treatment of focal hand dystonia. Front Hum Neurosci. 2015 Jul 9;9:385. doi: 10.3389/fnhum.2015.00385. eCollection 2015. PMID 26217209

RESULTS

PARTICIPANT FLOW:
Groups:
- rTMS + SMR, Then rTMS + CTL: Repetitive transcranial magnetic stimulation and sensorimotor retraining
  Repetitive Transcranial Magnetic Stimulation (Magstim): Applied to the premotor cortex at 1 Hz at 80% resting motor threshold for 1200 pulses.
  Sensorimotor Retraining: For sensorimotor retraining, a subset of the Learning-based Sensorimotor Training program was followed
- rTMS + CTL, Then rTMS + SMR: Repetitive transcranial magnetic stimulation (rTMS) with non-specific therapy that includes stretching, massage, range of motion
  Repetitive Transcranial Magnetic Stimulation (Magstim): Applied to the premotor cortex at 1 Hz at 80% resting motor threshold for 1200 pulses.
Period: Overall Study
Arm/Group | rTMS + SMR, Then rTMS + CTL | rTMS + CTL, Then rTMS + SMR
Started | 5 | 4
Completed | 4 | 4
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- rTMS + Sensorimotor Retraining, rTMS + CTL: Repetitive transcranial magnetic (rTMS) stimulation and sensorimotor retraining for the first phase, then rTMS with control therapy (CTL). CTL therapy was non-specific therapy that includes stretching, massage, range of motion.
  Repetitive Transcranial Magnetic Stimulation (Magstim): Applied to the premotor cortex at 1 Hz at 80% resting motor threshold for 1200 pulses.
  Sensorimotor Retraining: For sensorimotor retraining, a subset of the Learning-based Sensorimotor Training program was followed
- rTMS + CTL, rTMS + Sensorimotor Retraining: Repetitive transcranial magnetic stimulation (rTMS) with control therapy (CTL). CTL therapy was non-specific therapy that includes stretching, massage, range of motion for the first phase, then rTMS with sensorimotor retraining.
  Repetitive Transcranial Magnetic Stimulation (Magstim): Applied to the premotor cortex at 1 Hz at 80% resting motor threshold for 1200 pulses.
- Total: Total of all reporting groups
Arm/Group | rTMS + Sensorimotor Retraining, rTMS + CTL | rTMS + CTL, rTMS + Sensorimotor Retraining | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (13.55359731) | 44 (6.751543034) | 46 (10.64320336)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Global Rating of Change at Posttest (Day 5)
Description: Symptom severity was assessed using the global rating of change (GROC). For the GROC, participants were asked to identify between one to three functions most impacted by focal hand dystonia. At posttest 1 they were then asked to select a rating of perceived change that represented the level of function compared to baseline. Perceived change consisted of a ±7 point Likert scale (+7= a very great deal better, 0= no change, -7= a very great deal worse).
Time Frame: Baseline and Posttest
Population: All participants who completed the first phase were included in the analysis. Data were only analyzed in the first intervention period of the study because there was a lack of a washout effect between periods. This lack of washout made data from the second intervention period unreliable.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- rTMS With Sensorimotor Retraining: Repetitive transcranial magnetic stimulation and sensorimotor retraining
  Repetitive Transcranial Magnetic Stimulation (Magstim): Applied to the premotor cortex at 1 Hz at 80% resting motor threshold for 1200 pulses.
  Sensorimotor Retraining: For sensorimotor retraining, a subset of the Learning-based Sensorimotor Training program was followed
- rTMS With Control Therapy: Repetitive transcranial magnetic stimulation (rTMS) with non-specific therapy that includes stretching, massage, range of motion
  Repetitive Transcranial Magnetic Stimulation (Magstim): Applied to the premotor cortex at 1 Hz at 80% resting motor threshold for 1200 pulses.
Arm/Group | rTMS With Sensorimotor Retraining | rTMS With Control Therapy
Number analyzed (Participants) | 5 | 4
units on a scale | 1.3 [0 to 3] | 1.2 [-4 to 3]

2. Secondary Outcome: Change From Baseline in Arm Dystonia Disability Scale at Posttest (Day 5)
Description: The Arm Dystonia Disability Scale (ADDS) is a survey where participants rate task difficulty for activities such as writing, handling utensils, and buttoning on a scale of 1-4 (1 = no difficulty ,4 = not able or marked difficulty). This is a subjective assessment of impairment due to focal hand dystonia. Scores are determined using an equation: total points scored, divided by the maximum possible (23), multiplied by the quotient by 90 and subtract from 90%. Scores range from 0%-90% with higher scores indicating more function.
Time Frame: Baseline and Posttest
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of function
Arm/Group | rTMS With Sensorimotor Retraining | rTMS With Control Therapy
Number analyzed (Participants) | 5 | 4
percentage of function | 71.98 (7.031320694) | 71.42 (8.464086657)

3. Secondary Outcome: Change From Baseline in Sensation at Posttest (Day 5)
Description: Examinations included two point discrimination. Two-point discrimination threshold was completed using a Disk-Criminator™. Participants were asked to reply "one" or "two" after each presentation. Static and dynamic stimuli were presented to the index and ring fingers bilaterally, meaning it was presented as a static stimuli or it was slowly swept across the skin (dynamic).
Time Frame: Baseline and Posttest
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | rTMS With Sensorimotor Retraining | rTMS With Control Therapy
Number analyzed (Participants) | 5 | 4
Participants
  Improvement | 3 | 2
  No Change | 2 | 1
  Worsening | 0 | 1

4. Secondary Outcome: Change From Baseline in Cortical Silent Period at Posttest (Day 5)
Description: Cortical silent period (CSP) testing was completed during an isometric contraction of the target muscle whereby the motor evoked potential is followed by a short duration of electromyographic quiescence. The maximal voluntary contraction for finger abduction was recorded using a custom strain gauge placed around the index finger. Real-time visual feedback was given on a laptop screen to project the force produced by the participant and 20% of the maximum of three trials was calculated and displayed on a target line. For the CSP, participants were asked to contract until the target line was met, then a single transcranial magnetic stimulation pulse was delivered to the motor cortex. Ten trials were collected with a short rest period to prevent fatigue.
  CSP duration was calculated in milliseconds (ms). CSP EMG data were first rectified, and then a 10-ms moving average calculation was applied to the data. The onset of the CSP was set as the time point of the delivery of the TM
Time Frame: Baseline and Posttest
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | rTMS With Sensorimotor Retraining | rTMS With Control Therapy
Number analyzed (Participants) | 5 | 4
Participants
  Improvement | 2 | 1
  No Change | 2 | 1
  Worsening | 1 | 2

5. Secondary Outcome: Change From Baseline for Pressure During Hand Writing at Posttest (Day 5)
Description: Digitized handwriting was assessed using a computerized tablet (WACOM Co., Ltd., japan) with MovAlyzeR® (Neuroscript LLC, Tempe, AZ) hardware and software. Participants used a custom modified digitized pen (Kiko Software, Netherlands) to write in a self-selected pace and style on the tablet with real-time visual feedback. Writing tasks included "My country tis of thee" at a self-selected pace, repeated eight times. Data were sampled at 215 Hz (resolution: 5080 lpi, accuracy: ±0.01 pressure range: 0-800 g). Writing samples were segmented by points of minimal velocity into single strokes for analysis. Pressure for each stroke was automatically calculated within the software.
Time Frame: Baseline and Posttest
Population: One participant that did not display symptoms affecting handwriting and did not participate in the handwriting analysis. Data were only analyzed in the first intervention period of the study because there was a lack of a washout effect between periods. This lack of washout made data from the second intervention period unreliable.
Measure: Count of Participants; unit: Participants
Arm/Group | rTMS With Sensorimotor Retraining | rTMS With Control Therapy
Number analyzed (Participants) | 5 | 3
Participants
  Improvement | 2 | 2
  No Change | 3 | 1
  Worsening | 0 | 0

6. Secondary Outcome: Change From Baseline for Physician Rated Impairment at Posttest (Day 5)
Description: Video recordings were made as participants wrote on a pad of paper with pen. Participants were asked to draw a series of 10 loops across the pad of paper followed by "The dog is barking" and their signature, each repeated four times. A physician blinded to participant allocation rated recordings. Scoring criteria were adapted from a standardized writer's cramp rating scale (WCRS) (Wissel et al., 1996), rating pathological flexion or extension at the wrist, fingers and elbow, presence of tremor, dystonic posture, writing speed and latency of dystonic symptoms. Final scores are expressed as a rating listed as a movement score.
Time Frame: Baseline and Posttest
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | rTMS With Sensorimotor Retraining | rTMS With Control Therapy
Number analyzed (Participants) | 5 | 4
Participants
  Improvement | 2 | 0
  No Change | 3 | 3
  Worsening | 0 | 1

7. Secondary Outcome: Change From Baseline in Physical Function at Posttest (Day 5)
Description: Participants completed the full SF-36 assessment with subsection of interest: "physical functioning".
Time Frame: Baseline and Posttest
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | rTMS With Sensorimotor Retraining | rTMS With Control Therapy
Number analyzed (Participants) | 5 | 4
Participants
  Improvement | 1 | 0
  No Change | 4 | 2
  Worsening | 0 | 2

ADVERSE EVENTS:
Time Frame: Before and after each session of the intervention phase
Description: Participants were evaluated per-sequence due to the lack of washout effect. Each participant was asked to identify if an event occurred immediately after and the beginning of each session throughout the study. A list of common side-effects was presented to each participant to report 'yes or no' to each side effect.
Groups:
- rTMS With Sensorimotor Retraining, Then rTMS With CTL: Repetitive transcranial magnetic stimulation (rTMS) and sensorimotor retraining for first phase, then rTMS with control (CTL) therapy.
  Repetitive Transcranial Magnetic Stimulation (Magstim): Applied to the premotor cortex at 1 Hz at 80% resting motor threshold for 1200 pulses.
  Sensorimotor Retraining: For sensorimotor retraining, a subset of the Learning-based Sensorimotor Training program was followed
- rTMS With CTL, Then rTMS With Sensorimotor Retrain: Repetitive transcranial magnetic stimulation (rTMS) with control (CTL) non-specific therapy that includes stretching, massage, range of motion for first phase, then rTMS with sensorimotor retraining for second phase.
  Repetitive Transcranial Magnetic Stimulation (Magstim): Applied to the premotor cortex at 1 Hz at 80% resting motor threshold for 1200 pulses.
  Sensorimotor Retraining: For sensorimotor retraining, a subset of the Learning-based Sensorimotor Training program was followed
Arm/Group | rTMS With Sensorimotor Retraining, Then rTMS With CTL | rTMS With CTL, Then rTMS With Sensorimotor Retrain
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 3/5 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rTMS With Sensorimotor Retraining, Then rTMS With CTL (N=5) | rTMS With CTL, Then rTMS With Sensorimotor Retrain (N=4)
Headache (Nervous system disorders) | 0 (0) | 2 (8) — Mild headache sometimes accompanied by dizziness
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Abnormal Sleep Pattern (Psychiatric disorders) | 1 (2) | 0 (0)
Decreased balance (Nervous system disorders) | 2 (2) | 0 (0) — Feeling dizzy, off-balance
Mood change (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small sample size may have underpowered the study. The high variance seen in our single subject analysis is not unusual as a current conundrum in neuromodulation is the variable response between subjects to many different types of neuromodulation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes